CLINICAL TRIAL: NCT07228130
Title: Microrandomized Trial to Optimize Use of Burden-reducing Self-monitoring Approaches in Behavioral Obesity Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R01DK136216 (NIH); R01DK136216 (NIH)
Record Dates: First submitted 2025-11-11; First posted 2025-11-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Obesity & Overweight
Keywords: Online; Obesity; Weight Loss; Diet; Physical Activity
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: The interventional model is a micro-randomized trial, which involves sequential (within-subject) randomization to different self-monitoring approaches throughout behavioral obesity treatment. Each participant will receive a 24-week online behavioral obesity treatment program and will be randomized to one of five SM strategies every two weeks, resulting in a total of 12 randomizations per participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Online Behavioral Obesity Treatment with Full Dietary Self-monitoring (Experimental): The Online Behavioral Obesity Treatment intervention combined with the Full Dietary Self-monitoring intervention.
  Interventions: Behavioral: Online Behavioral Obesity Treatment; Behavioral: Full Dietary Self-monitoring
- Online Behavioral Obesity Treatment with Reduced-frequency Dietary Self-monitoring (Experimental): The Online Behavioral Obesity Treatment intervention combined with the Reduced-frequency Dietary Self-monitoring intervention.
  Interventions: Behavioral: Online Behavioral Obesity Treatment; Behavioral: Reduced-frequency Dietary Self-monitoring
- Online Behavioral Obesity Treatment with Self-Monitoring of Dietary Lapses Only (Experimental): The Online Behavioral Obesity Treatment intervention combined with the Self-Monitoring of Dietary Lapses Only intervention.
  Interventions: Behavioral: Online Behavioral Obesity Treatment; Behavioral: Self-Monitoring of Dietary Lapses Only
- Online Behavioral Obesity Treatment with Smartwatch-based Self-monitoring of Energy Intake (Experimental): The Online Behavioral Obesity Treatment intervention combined with the Smartwatch-based Self-monitoring of Energy Intake intervention.
  Interventions: Behavioral: Online Behavioral Obesity Treatment; Behavioral: Smartwatch-based Self-monitoring of Energy Intake
- Online Behavioral Obesity Treatment with Self-monitoring of Body Weight Only (Experimental): The Online Behavioral Obesity Treatment intervention combined with the Self-monitoring of Body Weight Only intervention.
  Interventions: Behavioral: Online Behavioral Obesity Treatment; Behavioral: Self-monitoring of Body Weight Only

INTERVENTIONS:
Behavioral: Online Behavioral Obesity Treatment — The online behavioral obesity treatment consists of: (a) 12 weekly multimedia lessons followed by 3 monthly lessons focused on behavioral skills for weight loss and weight loss maintenance; (b) online tools for goal setting, self-monitoring of diet, physical activity, and body weight; and (c) weekly feedback messages summarizing progress toward goals and providing support and problem-solving. Participants are given recommendations to help them set goals based on their self-monitoring condition (i.e., calorie goal, lapse goal, weight loss goal) and are guided to follow a healthy eating plan to achieve weight loss and health improvement. The physical activity goal is based on baseline activity level, with gradual progression from 50 minutes per week to 250 minutes per week of moderate-intensity activity (e.g., brisk walking).
  The program emphasizes evidence-based behavioral strategies including stimulus control, problem-solving, goal setting, and relapse prevention.
Behavioral: Full Dietary Self-monitoring — Recording all food and drink consumed, with calorie estimates, every day.
  Arms: Online Behavioral Obesity Treatment with Full Dietary Self-monitoring
Behavioral: Reduced-frequency Dietary Self-monitoring — Recording all food and drink consumed, with calorie estimates, on 3 days per week.
  Arms: Online Behavioral Obesity Treatment with Reduced-frequency Dietary Self-monitoring
Behavioral: Self-Monitoring of Dietary Lapses Only — Recording only episodes of eating or drinking that likely cause weight gain or put weight loss at risk.
  Arms: Online Behavioral Obesity Treatment with Self-Monitoring of Dietary Lapses Only
Behavioral: Smartwatch-based Self-monitoring of Energy Intake — Using a smartwatch that detects eating gestures and estimates energy intake (i.e., "calories") via built-in sensors.
  Arms: Online Behavioral Obesity Treatment with Smartwatch-based Self-monitoring of Energy Intake
Behavioral: Self-monitoring of Body Weight Only — Weighing daily using a smart scale that automatically syncs data to the online treatment platform.
  Arms: Online Behavioral Obesity Treatment with Self-monitoring of Body Weight Only

SUMMARY:
This clinical trial is focused on testing dietary self-monitoring strategies used in behavioral obesity treatment. The goal is to determine which self-monitoring strategies are most useful for whom, at which points in treatment, and under what circumstances.

Researchers will provide a 24-week online behavioral obesity treatment program, and will randomize participants to use one of 5 dietary self-monitoring strategies every two weeks. The five strategies include: recording all food and drink consumed and corresponding energy intake (i.e., "calories") on 7 days per week; recording all food and drink consumed and corresponding energy intake (i.e., "calories") on 3 days per week; self-monitoring of dietary lapses (i.e. any eating/drinking likely to cause weight gain or put weight loss at risk); smartwatch-based monitoring of energy intake (i.e., "calories"); and self-monitoring of body weight only via smart scale.

Participants will:

* Follow a 24-week online program for weight loss and health improvement
* Use the assigned self-monitoring strategy every two weeks
* Meet with the researchers periodically via online video call and provide research data by answering questions via periodic online surveys.

DETAILED DESCRIPTION:
This clinical trial is a 24-week micro-randomized trial (MRT) designed to optimize the use of dietary self-monitoring (SM) strategies during behavioral obesity treatment (BOT). Self-monitoring is considered the cornerstone of BOT because it enables individuals to regulate behaviors that influence energy balance and weight loss. However, adherence to traditional full dietary SM (i.e., recording all food and beverages consumed each day) declines rapidly over time due to its burden, leading to poorer weight loss outcomes.

To address this problem, this study evaluates five SM approaches that vary in intensity and burden:

1. Full dietary SM: Recording all food and drink consumed, with calorie estimates, every day.
2. Reduced-frequency dietary SM: Recording all food and drink consumed, with calorie estimates, on 3 days per week.
3. Self-monitoring of dietary lapses only: Recording only episodes of eating or drinking that likely cause weight gain or put weight loss at risk.
4. Smartwatch-based SM of energy intake: Using a smartwatch that detects eating gestures and estimates energy intake (i.e., "calories") via built-in sensors.
5. Body weight SM only: Weighing daily using a smart scale that automatically syncs data to the online treatment platform.

All participants (N=275 adults with overweight or obesity, aged 18-70) will receive a 24-week evidence-based, online BOT. This BOT includes interactive multimedia lessons on nutrition, physical activity, and behavioral skills for weight management, with individualized calorie and activity goals, self-regulation training, and automated feedback. The only experimental manipulation is the self-monitoring approach assigned every two weeks.

At the start of treatment and every two weeks thereafter, participants will be randomly assigned to one of the five SM approaches (12 total randomizations per participant). Randomization probabilities favor assignment to full dietary SM at treatment initiation, then gradually equalize across approaches. At each randomization, participants will be notified of their new SM assignment and receive a brief online training for that approach. A member of the research team will conduct a short online video call to confirm comprehension and assist with troubleshooting.

Participants will complete study assessments remotely at baseline and 24 weeks via online video call and online surveys. They will be provided with study equipment, including a smart scale and a smartwatch (participants may use their own smartwatch if it is compatible with the study platform). All SM data (e.g., SM logs, smartwatch data, smart scale readings) will be automatically transferred to the secure BOT system. Participants will also complete brief questionnaires at each randomization point assessing perceived burden, motivation, satisfaction, and engagement with the assigned SM approach.

The co-primary outcomes are (1) SM adherence, defined as the number of days per two-week period that the participant completes ≥2 eating recordings (or weighs daily in the body-weight-only condition), and (2) objectively measured weight change (kg) via smart scale. Secondary outcomes include perceived burden, motivation, satisfaction with SM strategy, and platform engagement metrics.

This MRT design enables the research team to compare short-term (2-week) effects of each SM approach on adherence and weight loss, identify how these effects vary over time and across individual characteristics, and develop a data-driven algorithm that adaptively selects optimal SM approaches for future treatment. Reinforcement learning will be applied to the MRT data to construct an adaptive SM-selection algorithm capable of personalizing SM recommendations based on individual differences, social determinants of health, and ongoing treatment response.

This project will yield both broadly applicable recommendations (e.g., which SM approaches are generally most effective at different stages of treatment) and an adaptive algorithm to guide individualized SM strategies in future clinical and research settings. The findings are expected to enhance long-term adherence to self-monitoring and improve the effectiveness and scalability of behavioral obesity treatments delivered online.

ELIGIBILITY:
* English language fluent and literate at the 6th grade level
* Body mass index (BMI) above 25 kg/m-squared
* Able to walk 2 city blocks without stopping
* Not currently participating in another weight loss program
* Not currently taking weight loss medication
* Has not lost ≥5% of body weight in the 6 months prior to enrolling
* Has not been pregnant within the 6 months prior to enrolling
* Does not plan to become pregnant within 12 months of enrolling
* Denies having a heart condition, chest pain during periods of activity or rest, or loss of consciousness in the 12 months prior to enrolling
* Denies any medical condition that would affect the safety of participating in unsupervised physical activity
* Denies any condition that would result in inability to follow the study protocol, including terminal illness, substance abuse, eating disorder (not including Binge Eating Disorder) and untreated major psychiatric illness
* Owns a smartphone compatible with study procedures and is willing to use it for study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to Self-Monitoring | 24 weeks
  Number of days on which the assigned self-monitoring strategy was used
Weight Change | 24 weeks
  Weight measured in kg on the provided home scale

SECONDARY OUTCOMES:
Perceived Burden of Assigned Self-Monitoring Approach | 24 weeks
  Self-reported perceived burden of the self-monitoring approach used during the prior 2 weeks, assessed with items adapted from the User Burden Scale (e.g., "Using this self-monitoring method required too much mental effort"). Higher scores indicate greater perceived burden.
Motivation to Engage in Self-Monitoring | 24 weeks
  Self-reported motivation to adhere to the assigned SM approach, measured using adapted items from the Motivation for Weight Loss Scale (e.g., "I intend to self-monitor using the assigned strategy on most days over the next two weeks").
Satisfaction With Assigned Self-Monitoring Approach | 24 weeks
  Self-reported satisfaction with the assigned SM strategy, assessed using items adapted from the Diabetes Treatment Satisfaction Questionnaire (e.g., "How satisfied were you with this self-monitoring strategy?").

CONTACTS AND LOCATIONS:
Overall Officials: Graham Thomas, PhD, Principal Investigator — The Miriam Hospital; Stephanie Goldstein, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Weight Control and Diabetes Research Center of The Miriam Hospital & Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified baseline data collected via online questionnaire, co-primary outcomes (i.e., participant adherence to SM conditions and weekly weights), data collected via the obesity treatment platform (e.g., website engagement), and data on treatment factors collected at 2-week intervals via questionnaire (e.g., perceived burden, satisfaction) will be shared with participants' consent. Identifiable and quasi-identifiable information will not be shared . Analyzed datasets along with analysis code and codebooks will be preserved and shared. Data will be made accessible via online repository at the time of associated publication(s) or the end of the performance period, whichever comes first, and they will remain publicly accessible as long as it is anticipated that they are useful for the larger research community, institutions, and/or broader public (to be determined by NIDDK-CR or VIVLI protocol).